CLINICAL TRIAL: NCT05131061
Title: 68Ga-Pentixafor PET/CT for the Subtyping Diagnosis of Primary Aldosteronism: A Prospective Diagnostic Accuracy Study
Brief Title: 68Ga-Pentixafor PET/CT for the Subtyping Diagnosis of Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Qifu Li (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2021-553
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Primary Aldosteronism
Keywords: PET CT; Primary aldosteronism; Adrenal venous sampling
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fasting plasma were collected for each patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unilateral primary aldosteronism(UPA): PA confirmatory tests was positive; successful intubation (SI ≥ 3) and LI ≥ 4; If LI between 2 and 4, should be combined with contralateral inhibition index < 1 or CT indicate typical adenomas on the dominant side.
  Interventions: Diagnostic Test: 68Ga-Pentixafor PET/CT imaging
- bilateral adrenal hyperplasia(BAH): PA confirmatory tests was positive; successful intubation (SI ≥ 3) and LI < 2; or LI between 2 and 4 but does not meet the UPA conditions
  Interventions: Diagnostic Test: 68Ga-Pentixafor PET/CT imaging

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor PET/CT imaging — 68Ga-Pentixafor PET/CT imaging

SUMMARY:
To evaluate the value of 68Ga-Pentixafor PET/CT in the diagnosis of primary aldosteronism subtype

DETAILED DESCRIPTION:
This is a prospective study. We will enroll 100 patients with definite diagnosis of PA using adrenal venous sampling(AVS) as the gold standard for subtype to evaluate the value of 68Ga-pentixaforPET/CT in the diagnosis of PA.

ELIGIBILITY:
Inclusion Criteria:

1. PA diagnosis confirmed by at least one confirmatory test
2. willingness to undergo AVS and surgery
3. informed consent to participate in the study.

Exclusion Criteria:

1. PA patients who met guideline criteria for bypassing AVS [i.e. younger than 35 years old, with typical APA characteristics (plasma aldosterone >300pg/ml, plasma renin < 2·5mIU/l, serum potassium <3·5mmol/l, CT indicated unilateral 1cm low-density adenoma);
2. failed adrenal vein cannulation during AVS;
3. Subtyping diagnosis was inconclusive based on AVS results (e.g. aldosterone/cortisol ratio in bilateral adrenal veins lower than the peripheral vein, or missing data);
4. pregnant or lactating women;
5. patients with a history of uncontrolled malignant tumor;
6. concurrent Cushing's syndrome [including mild autonomous cortisol secretion: cortisol after 1mg dexamethasone suppression test (DST)>138 nmol/l or cortisol after 2mg DST >50 nmol/l or cortisol after 1mg DST 50-138 nmol/l plus adrenocorticotrophic hormone (ACTH)<10pg/ml;
7. diagnosis of familial hyperaldosteronism;
8. imaging characteristics suggestive of pheochromocytoma or adrenal cortical carcinoma;
9. unsuitable for surgery, such as heart failure with New York Heart Association (NYHA) class III or IV, severe anemia (Hemoglobin<60g/L), stroke or acute coronary syndrome within 3 months, severe ascites and cirrhosis, estimated glomerulus filtration rate<30ml/min/m;
10. alcohol or drug abuse and mental disorders.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Power Analysis and Sample Size software 11 (PASS 11) was used to calculate the sample size. A sample of 40 from the positive group (i.e. UPA group) and 60 from the negative group (i.e. BPA group) achieves 84% power to detect a difference of 0·15 between the area under the receiver-operator characteristics curve (AUC) under the null hypothesis of 0·70 and an AUC under the alternative hypothesis of 0·85 using a two-sided z-test at a significance level of 0·05.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
accuracy of 68Ga-PentixaforPET/CT in subtyping diagnosis of PA | at the end of study(the last enrolled patient completed a 3-month follow-up)
  AUC

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Mulatero P, Sechi LA, Williams TA, Lenders JWM, Reincke M, Satoh F, Januszewicz A, Naruse M, Doumas M, Veglio F, Wu VC, Widimsky J. Subtype diagnosis, treatment, complications and outcomes of primary aldosteronism and future direction of research: a position statement and consensus of the Working Group on Endocrine Hypertension of the European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1929-1936. doi: 10.1097/HJH.0000000000002520. PMID 32890265
- [Result] Young WF, Stanson AW, Thompson GB, Grant CS, Farley DR, van Heerden JA. Role for adrenal venous sampling in primary aldosteronism. Surgery. 2004 Dec;136(6):1227-35. doi: 10.1016/j.surg.2004.06.051. PMID 15657580
- [Result] Rossi GP, Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J Jr, Naruse M, Deinum J, Schultze Kool L, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Christian Rump L, Vonend O, Willenberg HS, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Dun Wu K, Wu VC, Kratka Z, Barbiero G, Battistel M, Chang CC, Vanderriele PE, Pessina AC. Clinical Outcomes of 1625 Patients With Primary Aldosteronism Subtyped With Adrenal Vein Sampling. Hypertension. 2019 Oct;74(4):800-808. doi: 10.1161/HYPERTENSIONAHA.119.13463. Epub 2019 Sep 3. PMID 31476901
- [Result] Kempers MJ, Lenders JW, van Outheusden L, van der Wilt GJ, Schultze Kool LJ, Hermus AR, Deinum J. Systematic review: diagnostic procedures to differentiate unilateral from bilateral adrenal abnormality in primary aldosteronism. Ann Intern Med. 2009 Sep 1;151(5):329-37. doi: 10.7326/0003-4819-151-5-200909010-00007. PMID 19721021
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Amar L, Baguet JP, Bardet S, Chaffanjon P, Chamontin B, Douillard C, Durieux P, Girerd X, Gosse P, Hernigou A, Herpin D, Houillier P, Jeunemaitre X, Joffre F, Kraimps JL, Lefebvre H, Menegaux F, Mounier-Vehier C, Nussberger J, Pagny JY, Pechere A, Plouin PF, Reznik Y, Steichen O, Tabarin A, Zennaro MC, Zinzindohoue F, Chabre O. SFE/SFHTA/AFCE primary aldosteronism consensus: Introduction and handbook. Ann Endocrinol (Paris). 2016 Jul;77(3):179-86. doi: 10.1016/j.ando.2016.05.001. Epub 2016 Jun 15. PMID 27315757
- [Result] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316
- [Result] Ding J, Zhang Y, Wen J, Zhang H, Wang H, Luo Y, Pan Q, Zhu W, Wang X, Yao S, Kreissl MC, Hacker M, Tong A, Huo L, Li X. Imaging CXCR4 expression in patients with suspected primary hyperaldosteronism. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2656-2665. doi: 10.1007/s00259-020-04722-0. Epub 2020 Mar 23. PMID 32206838